CLINICAL TRIAL: NCT03130998
Title: A Cluster Randomized Trial of Tailored vs Generic Knowledge Brokering to Integrate Mood Management Into Smoking Cessation Interventions in Primary Care Settings in Ontario, Canada
Brief Title: Cluster Randomized Trial of Knowledge Brokering to Integrate Mood and Smoking Cessation in Ontario Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Peter Selby, Director, Medical Education, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 065-2016
Record Dates: First submitted 2017-04-18; First posted 2017-04-27 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Depression
Keywords: smoking cessation; depression; mental health; mood management; primary care; screening; brief intervention; referral to treatment
MeSH Terms: conditions — Depression; Smoking Cessation; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study design is a cluster (cluster = clinical practice) randomized trial of FHTs participating in the STOP program. FHTs in the STOP program will be randomly allocated 1:1 to receive either generalized messages (related to depression and smoking) exclusively via email (Group A) or be assigned an eKB who provides personalized support through phone- and email-based check-ins (Group B). Academic affiliation and cluster size will be treated as balancing factors in a stratified allocation or as covariates in the statistical analyses.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Group A (Active Comparator): When a patient is screened as showing depressive symptoms, the practitioner will be prompted to intervene and refer that patient to treatment. The practitioner will receive knowledge broker support to carry out these actions in the form of one email per month for one year. The first email will provide an electronic copy of a Cochrane review (describing the link between smoking and mood) and a short description of the integration of a depression ICP in the STOP portal. The STOP YouTube channel with detailed instructions on how to use the revised portal will be made available. Subsequent communications will be based on general needs identified at baseline and content discussed in the STOP Community of Practice (teleconferences, online forum between STOP practitioners).
  Interventions: Behavioral: Emails
- Intervention - Group B (Experimental): When a patient is screened as showing depressive symptoms, the practitioner will be prompted to intervene and refer that patient to treatment. The practitioner will receive individualized support through a remote knowledge broker (rKB) communicating via interactive technology. The rKB will be certified in tobacco cessation counseling through CAMH's TEACH program and will have completed a specialty course on tobacco addiction treatment in those with mental illness. The rKB will have access to the CAMH network of KBs (e.g. Evidence Exchange Network ) for guidance and support, as this has been shown to be important for KB success.
  Interventions: Behavioral: Remote Knowledge Broker (rKB)

INTERVENTIONS:
Behavioral: Remote Knowledge Broker (rKB) — The intervention is the tailored support received by a knowledge broker via technology in Group B. The rKB will: ensure relevant research evidence related to depression and smoking is transferred to the FHTs in ways that are most useful to them; develop capacity for evidence-informed decision-making at each site; and assist sites in translating evidence into local practice. These tasks will be accomplished by an initial 2-hour, virtual visit with each site and regular phone- and email-based check-ins. The specific tasks will be dictated by the needs of each site, and will create opportunity for practitioners to share their experiences with the rKB, learn new evidence, and work with the rKB on how to best implement the evidence.
  Arms: Intervention - Group B
Behavioral: Emails — When a patient is screened as showing depressive symptoms, the practitioner will be prompted to intervene and refer that patient to treatment. The practitioner will receive knowledge broker support to carry out these actions in the form of one email per month for one year. The first email will provide an electronic copy of a Cochrane review (describing the link between smoking and mood) and a short description of the integration of a depression ICP in the STOP portal. The STOP YouTube channel with detailed instructions on how to use the revised portal will be made available. Subsequent communications will be based on general needs identified at baseline and content discussed in the STOP Community of Practice (teleconferences, online forum between STOP practitioners).
  Arms: Control - Group A

SUMMARY:
Compared to smokers who are not depressed, smokers with depression who try to quit smoking are 10% less likely to succeed when given standard treatment. A simple program with a detailed handout on relaxation exercises and a journal to record mood and urges to smoke when trying to quit has been shown to increase quit success in depressed smokers by 12 to 20%. However, it remains unclear how to best implement this knowledge into primary care settings.

Through this study, the investigators will seek to answer the following questions:

* Does a knowledge broker communicating via generic email reminders engage clinicians to provide patients resources for mood management more or less frequently than via interactive technology (eKB)?
* Which Knowledge Translation (KT) strategy used to change clinicians' behavior (emails vs. eKB) has the greatest effect on smoking quit rates in depressed smokers?
* What is the incremental cost effectiveness of the two KT strategies?

DETAILED DESCRIPTION:
Given the cost-effectiveness of smoking cessation programs, the Centre for Addiction and Mental Health implemented the STOP program in 147 Family Health Teams (FHTs) treating 47,888 smokers with nicotine replacement therapy and counselling. Following the knowledge to action framework every FHT in STOP uses a web portal with an integrated decision aid, data collection, and feedback tool. Though STOP data finds lower quit rates among smokers with depression, it currently does not offer specialized clinical pathways for depressed smokers.

Both smoking and depression are major public health problems with high morbidity and mortality. Individuals with depression are almost twice as likely to be smokers, have lower long-term smoking abstinence (OR=0.81, 95% CI=0.67-0.97), and experience greater addiction severity and negative mood when quitting smoking. In the STOP Program, 38% of smokers have current or past depression; their 6-month quit rates are significantly lower than participants without depression (33% vs. 40%, p<0.001). This has led FHT-STOP practitioners to express the need for specialized clinical pathways for depressed smokers.

Self-help mood management (relaxation exercises and mood monitoring) integrated with smoking cessation treatment increases long-term quit rates by 12 to 20%. More research is needed to test the effectiveness of an integrated care pathway (ICP) for depression as part of cessation treatment. It is unclear which KT strategy would be more effective in engaging clinicians and driving behavior change. A randomized controlled trial in Public Health Units (PHUs) found no difference in health care provider behavior when prompted by a knowledge broker, emails or websites. However , similar to other studies, it showed the need to match organizational research culture to KT strategy; emails worked better in PHUs with a strong research culture, while KBs seemed more suitable in PHUs where research culture was low. Given that FHTs range anywhere from academic- to community-based research cultures, it is unclear which KT strategy will be most effective.

CAMH's existing Smoking Treatment for Ontario Patients (STOP) program works in partnership with 80% of eligible Family Health Teams (FHTs) in Ontario and has treated 47,888 smokers with free nicotine replacement and counselling since July 2011. Based on data already collected in the STOP Program, the STOP portal (an online data management and collection tool used by all STOP practitioners to complete participant enrollment and record smoking status at each visit), will flag smokers with current or past depressive symptoms. FHTs will be randomly allocated 1:1 to receive messages regarding depression and smoking exclusively via email (Group A) or via an eKB who will develop a one-on-one relationship with clinicians through frequent phone calls, web conferencing, and emails (Group B). The investigators will compare which method is more effective in changing clinician behavior by recording the number of times resources are provided to eligible patients. Investigators will also compare the smoking quit rates of patients from the two groups at 6-month follow-up and ask clinicians and patients what they liked and disliked about the program.

ELIGIBILITY:
Inclusion Criteria:

* Must be Family Health Team (FHT) participating in the Smoking Treatment for Ontario Patients (STOP) program
* FHT must use online portal to complete STOP questionnaires, in English, in real-time with patient

Exclusion Criteria:

* Non-FHTs participating in STOP program
* Clinics who conduct STOP questionnaires exclusively on paper, or in French, or not in real-time with patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2765 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Resource accepted by patient | : Approximately 2-5 minutes as part of a brief intervention between the practitioner and patient
  The primary outcome will be the provision of the mood management intervention to eligible patients upon completion of the STOP smoking cessation program enrollment. This dichotomous outcome will be measured as positive by a response of "Patient accepted the resource" to the practitioner question "Did the patient accept or decline the resource?". In contrast, the outcome will be measured as negative if given a response of "Patient declined the resource" to the practitioner question "Did the patient accept or decline the resource?" or a response of "no" to the practitioner directive "Provide this patient with resources on mood management."

SECONDARY OUTCOMES:
Smoking Abstinence | Approximately 10 minutes during 1-hour appointment between practitioner and patient
  The secondary outcome, measured at the site level, is the proportion of eligible baseline visits which result in practitioners delivering the mood management intervention to patients as measured by the STOP Portal system (patient accepts practitioner's offer of intervention).
Cost-effectiveness | 6-month follow-up
  The tertiary outcome will be a cost-effectiveness analysis (CEA), evaluating the delivery of each intervention from the health care system, and societal perspectives. The CEA will include the costs of developing, maintaining, and running each intervention in addition to costs associated with personnel, training, supplies, and services. The incremental cost-effectiveness ratio (ICER) will be the primary outcome of the CEA. An additional measure of interest will be the 95% confidence interval for the ICER
Decrease in depression scores | 6-month follow-up
  Other outcomes measured in this study will include change in The Patient Health Questionnaire (PHQ)-9 score between the baseline and 6-month follow-up surveys. Scores in the PHQ-9 range from 0-27; the higher the score the more likely the person has more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, MBBS CCFP FCFP MHSc DipABAM, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minian N, Noormohamed A, Baliunas D, Zawertailo L, Mulder C, Ravindran A, de Oliveira C, Selby P. Tailored Versus Generic Knowledge Brokering to Integrate Mood Management Into Smoking Cessation Interventions in Primary Care Settings: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2018 Apr 27;7(4):e111. doi: 10.2196/resprot.9715. PMID 29703714
- [Derived] Minian N, Ahad S, Ivanova A, Veldhuizen S, Zawertailo L, Ravindran A, de Oliveira C, Baliunas D, Mulder C, Bolbocean C, Selby P. The effectiveness of generic emails versus a remote knowledge broker to integrate mood management into a smoking cessation programme in team-based primary care: a cluster randomised trial. Implement Sci. 2021 Mar 20;16(1):30. doi: 10.1186/s13012-021-01091-6. PMID 33743777